CLINICAL TRIAL: NCT03407287
Title: Peripheral Venous Analysis (PIVA) for Predicting Volume Responsiveness and Fluid Status:
Brief Title: Peripheral Venous Analysis (PIVA) for Predicting Volume Responsiveness and Fluid Status
Acronym: PIVA
Status: Terminated | Type: Observational
Why Stopped: interim analysis, closed for additional product development
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Kelly Kohorst, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: 828397
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Systemic Inflammatory Response Syndrome; Distributive Shock; Hypotension and Shock; Decompensated Congestive Heart Failure; Atrial Fibrillation; High Risk Non-cardiac Surgery
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Hypotension; Shock; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Cardiac Catheterization
  Interventions: Procedure: Peripheral Intravenous Analysis (PIVA); Procedure: Standard of care invasive vascular monitoring; Procedure: Standard noninvasive vascular monitoring
- Distributive shock
  Interventions: Procedure: Peripheral Intravenous Analysis (PIVA); Procedure: Standard of care invasive vascular monitoring; Procedure: Standard noninvasive vascular monitoring
- Vasoactive and inotropic agents
  Interventions: Procedure: Peripheral Intravenous Analysis (PIVA); Procedure: Standard of care invasive vascular monitoring; Procedure: Standard noninvasive vascular monitoring
- Congestive heart failure
  Interventions: Procedure: Peripheral Intravenous Analysis (PIVA); Procedure: Standard of care invasive vascular monitoring; Procedure: Standard noninvasive vascular monitoring
- Atrial fibrillation: Patients with atrial fibrillation undergoing elective direct current cardioversion
  Interventions: Procedure: Peripheral Intravenous Analysis (PIVA); Procedure: Standard of care invasive vascular monitoring; Procedure: Standard noninvasive vascular monitoring
- Patients undergoing surgery: Patients undergoing surgery requiring positive pressure ventilation and arterial line placement
  Interventions: Procedure: Peripheral Intravenous Analysis (PIVA); Procedure: Standard of care invasive vascular monitoring; Procedure: Standard noninvasive vascular monitoring

INTERVENTIONS:
Procedure: Peripheral Intravenous Analysis (PIVA) — Non-invasive measurement of peripheral venous waveform analysis (PIVA) obtained by connecting a standard transducer (AD Instruments, Colorado Springs, Co) to a universal adaptor or stopcock on a peripheral IV
Procedure: Standard of care invasive vascular monitoring — Standard of care invasive monitoring in the intensive care settings with central venous catheters, pulmonary artery catheters, or trans-esophageal echocardiography for determining volume status.
Procedure: Standard noninvasive vascular monitoring — Standard noninvasive vascular monitoring of blood pressure, pulse rate, pulse oximetry and respiratory rate.

SUMMARY:
The aim of this study is to determine the effects of fluid alternations, hemodynamic changes, mechanical ventilation, pharmacologic agents, positional changes, and comorbidities on the Peripheral Intravenous waveform Analysis (PIVA) signal.

DETAILED DESCRIPTION:
Intravascular volume status determination remains elusive. Standard vital sign monitoring, including heart rate and blood pressure, fails to detect intravascular volume depletion and volume overload. Likewise, invasive monitoring is fraught with risk including vascular injury and central line associated infections. As such, a minimally-invasive mechanism to overcome the barriers of standard monitoring to detect volume status derangement, would be highly valuable. The goal of the study is to perform a series of observational feasibility studies in healthy and hospitalized subjects to determine effects of fluid alternations, hemodynamic changes, mechanical ventilation, pharmacologic agents, positional changes, and comorbidities on the PIVA signal

ELIGIBILITY:
Cardiac Catheterization

Inclusion criteria:

* Patients undergoing right heart catheterization or left and right heart catheterizaton; Age >=18

Exclusion criteria:

* Cardiac assist devices (intra-aortic balloon pump, ventricular assist devices, and extra corporeal membrane oxygenation), ongoing ACLS, aortic or mitral valve disease greater than mild in severity, aortic or mitral valve replacement, active irregular heart rhythm, patients with restrictive cardiomyopathies (cardiac amyloidosis), constrictive cardiac disease (constrictive pericarditis or cardiac-tamponade), congenital heart disease other than foramen ovale, repaired atrial or ventricular septal defect, female patients who are pregnant or lactating, or patients with known psychiatric or neurological disease who are unable to consent. Patients who do not have a functional peripheral IV as part of standard care. Pressors, starches, lipids, propofol, or D10 or higher running through the PIVA line.

Distributive Shock

Inclusion Criteria:

* Cardiopulmonary bypass for cardiac procedures within one hour of arriving in the ICU post-op; Age >=18

Exclusion Criteria:

* Cardiac assist devices (intra-aortic balloon pump, ventricular assist devices, and extracorporeal membrane oxygenation), ongoing ACLS, severe tricuspid regurgitation or stenosis, patient with restrictive cardiomyopathies (cardiac amyloidosis), patients receiving pulmonary vasodilators (nitric oxide, sodium nitroprusside, sildenafil), atrial fibrillation, congenital heart disease, female patients who are pregnant or lactating, or patients with known psychiatric or neurological disease who are unable to consent. Patients who do not have a functional peripheral IV as part of standard care.

Vasoactive and Inotropic Agents

Inclusion Criteria:

* Hospitalized patients with central venous access and pulmonary arterial catheter in place, requiring infusion of vasoactive and/or inotropic agents; Age >=18

Exclusion Criteria:

* Cardiac assist devices (intra-aortic balloon pump, ventricular assist devices, and extracorporeal membrane oxygenation), ongoing ACLS, severe tricuspid regurgitation or stenosis, patient with restrictive cardiomyopathies (cardiac amyloidosis), patients receiving pulmonary vasodilators (nitric oxide, sodium nitroprusside, sildenafil), atrial fibrillation, congenital heart disease, female patients who are pregnant or lactating, or patients with known psychiatric or neurological disease who are unable to consent. Patients who do not have a functional peripheral IV as part of standard care.

Congestive Heart Failure

Inclusion Criteria:

* Patients presenting to Vanderbilt University Medical Center with the diagnosis of congestive heart failure and present with symptoms of fluid overload; Age>=18

Exclusion Criteria:

* Cardiac assist devices (intra-aortic balloon pump, ventricular assist devices, and extra corporeal membrane oxygenation), ongoing ACLS, active irregular heart rhythm, patient with restrictive cardiomyopathies (cardiac amyloidosis), or constrictive cardiac disease (constrictive pericarditis or cardiac tamponade), congenital heart disease other than foramen ovale, repaired atrial or ventricular septal defect, female patients who are pregnant or lactating, or patients with known psychiatric or neurological disease who are unable to consent. Patients who do not have a functional peripheral IV as part of standard care.

Atrial Fibrillation (undergoing elective direct current cardio version)

Inclusion Criteria:

* Patients with atrial fibrillation undergoing direct current cardioversion; Age >=18

Exclusion Criteria:

* Cardiac assist devices (intra-aortic balloon pump, ventricular assist devices, and extra corporeal membrane oxygenation), ongoing ACLS, patients with restrictive cardiomyopathies (cardiac amyloidosis) or constrictive cardiac disease (constrictive pericarditis or cardiac tamponade), congenital heart disease other than foramen ovale, repaired atrial or ventricular septal defect, female patients who are pregnant or lactating, or patients with known psychiatric or neurological disease who are unable to consent. Patients who do not have a functional peripheral IV as part of standard care.

Patients undergoing Surgery

Inclusion Criteria:

* Patients presenting for surgery requiring positive pressure ventilation and arterial line placement; Age >=18

Exclusion Criteria:

* Cardiac assist devices (intra-aortic balloon pump, ventricular assist devices, and extra corporeal membrane oxygenation), ongoing ACLS, patients with restrictive cardiomyopathies (cardiac amyloidosis) or constrictive cardiac disease (constrictive pericarditis or cardiac tamponade), active irregular cardiac rhythm, congenital heart disease other than foramen ovale , repaired atrial or ventricular septal defect, female patients who are pregnant or lactating, patients with known psychiatric or neurological disease who are unable to consent, or any other medical condition which, in the opinion of the investigator, would place the patient at undue risk from participation in the trial. Patients who do not have a functional peripheral IV as part of standard care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients hospitalized at Vanderbilt University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Correlation of PIVA score to standard hemodynamic monitors | Baseline to end of monitoring (Approximately 180 minutes)
  Peripheral intravenous waveform analysis score is used to detect intravascular volume status. The scale ranges from 2-40 and is interpreted as a surrogate for pulmonary capillary wedge pressure. The normal scale range is 6-12. A PIVA score of 2 indicates a low intravascular volume and 40 indicates a high intravascular volume.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly L. Kohorst, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No